CLINICAL TRIAL: NCT06127680
Title: Feasibility Study to Test the Implementation of Health Promotion Advice (Exercise and Protein Intake) for Older People Attending a Community Mental Health Service.
Brief Title: Brief Health Promotion Intervention for Older People in Mental Health
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Corina Naughton, Professor Corina Naughton, University College Cork
Other Study IDs: ECM 4 (w) 14/02/2023
Record Dates: First submitted 2023-09-25; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue; Frailty
Keywords: Mental health; Older People; Health promotion; Exercise; Nutrition; Frailty
MeSH Terms: conditions — Frailty; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Brief Health Promotion Advice — Brief Health Promotion advice on exercise and nutrition (protein intake) delivered by a health care professional during routine consultations

SUMMARY:
The goal of this observational study is to test the delivery of brief health promotion advice with supporting information leaflets as part of standard clinical consultation for older people attending a community mental health service

The main questions it aims to answer are:

1. Is a brief health promotion intervention designed for primary care transferable and acceptable to older people attending acute community-based mental health services (Travers et al 2022)
2. Can older adults with ongoing mental health conditions be recruited and retained in the study
3. Will participants adhere to the health promotion intervention over a three-month period
4. Can evaluation data be collected from participants

Eligible participants will be asked to:

* participate in a brief health promotion (10 minutes) advice given by an advanced nurse practitioner (ANP) in mental health during a routine outpatient clinic/home visit
* participants receive exercise and protein advice leaflets (laminated)
* participants rehearse the exercise with the ANP
* one-month follow-up by ANP to assess and promote adherence to the intervention Researchers will use a one-group pre-post test study to compare baseline data on physical and mental health outcomes to participants' outcomes at three-month follow-up (there is no control group).

DETAILED DESCRIPTION:
Target Population

The target population is older adults attending mental health services aged 65 years and older. Age 65 years is the age for referral to older adult mental health services. The Older adult mental health services provide care and treatment for people aged over 65's who develop new onset functional mental illnesses such as depression, and severe anxiety or those with a diagnosis of dementia with behavioural and psychological problems requiring specialist intervention and care.

In the feasibility study Sample size, the aim is to recruit 15-20 patients to test the feasibility of the intervention in this population.

Study Design

The study will be a one-group pretest -posttest intervention design with a patient survey at baseline, 1-month and 3-month follow-up. The project will be undertaken over 12 months. Once ethical approval is obtained, patient recruitment and baseline data will be collected and the intervention will be delivered: in March - June 2023, 1 month follow-up April to July and three month follow-up August to October 2023.

Data Collection The ANP will complete the structured questionnaire with the patient in the MH clinic or patient home during routine clinical consultations. The one-month and three month follow-up will be via telephone or in the OPD clinic/persons' home as part of normal schedule of visits. No extra clinic or home visits are planned as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* For the purpose of this study service users eligible for the study are:

  1. Aged 65 years and older
  2. Cognitive capacity to provide informed consent
  3. Attending Older adult mental health services
  4. Mental Health team deem the client stable and able to participate in the intervention
  5. Patient independently mobile and living in the community (may use a walk aid)(Clinical Frailty Scale ≤5)

     Exclusion Criteria:

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: 1. Service users with moderate advanced dementia will be excluded as the intervention is unsupervised.
  2. Patents that cannot provide informed consent
  3. Patients who cannot understand English or require a translator
  4. Patients experience acute mental health crisis
  5. Patients with significant restricted mobility, using Zimmer frame inside or outside their house (CFS≥5)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
SARC-F (tool title not an abbreviation) | Baseline 3-month follow-up
  The SARC-F is a screening tool for sarcopenia (Malmstrom et al 2013). SARC-F comprises five components using self-report on: strength, assistance walking, rise from a chair, climb stairs, and falls. SARC-F scale scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst) and are dichotomized to represent symptomatic (4+) vs. healthy (0-3) status (Malmstrom et al 2016).

SECONDARY OUTCOMES:
Clinical Frailty Scale | Baseline and 3 months
  Clinical Frailty Scale (CSF) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill), a higher score indicates poorer physical and cognitive function (Rockwood et al 2005, Church 2020).
Global Physical Health Scale (GPHS) V1.2 | Baseline and 3 months
  The Global Physical Health Scale v1.2 is a four-item validated general health questionnaire Riley et al 2010, Hays et al 2015). Four items are used to assess global physical health. Three items (rate your physical health, everyday activities , rate your fatigue ) of these are administered using five-category response scales. Higher scores indicated better health. One item (rating of pain on average) uses a response scale of 0-10 that is recoded to five categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5), the scale is then reverse coded, i.e. 0 (no pain)= 5). Overall scores range from 5 to 20 indicating best possible physical health (PROMIS 2021)
Mental wellbeing (bespoke items) | Baseline and 3 months
  Two items (rate your overall mental health, rate your mood/ sense of well-being) over past seven days was rated on a 5 point scale (excellent =5; very poor =1). Higher score indicates better mental health. Items are not combined for overall score
Yale Physical Assessment Scale | Baseline and 3 months
  Two items from Yale Physical Assessment Scale (vigorous exercise frequency and duration over past 7 days, and Walking for exercise frequency and duration over past 7 days ((De Abajo et al., 2001). Frequency was rated on a 4 point scale (not at all=0; 1-2 times=1, 3-4 times=2 or >4 times=3) Duration (0=not applicable, 1=10-30 mins, 2=31-60 mins, 3> 60 mins. Scores are calculated by multiplying Frequency score X Duration score (no weight was applied). Higher scores indicate more activity. Items were not combined for an overall exercise score.
  Post intervention, we added an additional question specific to the exercises on the information leaflet In the past week (7 days) have you completed the exercises on the information leaflet Frequency (None=0, 1 day=1, 2 days=2; 3 days=3, 4days=4, 5 days=5); X Duration (none =0; 10 mins=1, 11-20 mins=2 , 21-30 mins=3, >30 mins=4). Higher values indicate greater exercise intensity (min score 0 to 20).
Simplified nutritional appetite questionnaire (SNAQ) | Baseline and 3 months
  questionnaire (SNAQ) is a four item scale (rate appetite, When I eat I feel full, food tastes, normally I eat) are rated on a five point scale (1 to 5). Total possible score range from 5 to 20, higher scores indicate better appetite. SNAQ score 14 indicates significant risk of at least 5% weight loss within six months (Kruizenga et al., 2005).
Protein intake | Baseline and 3 months
  Self-report number of protein portions eaten on previous day. Protein was categorised as: meat/fish; milk/diary; eggs/cheese; vegetable protein

OTHER OUTCOMES:
Acceptability (Bespoke item) | 1 and 3 month follow-up
  One item measures acceptability: The exercise and nutrition advice was acceptable to me (made sense) rated on a 5 point Likert scale (1=strongly disagree to 5 strongly agree)
Ease of Use (Bespoke item) | 1 and 3 month follow-up
  One item measured Ease of Use ' To what extent was it easy to incorporate the exercise an nutrition advice into your daily routine rated on a five point Likert scale (1=very difficult to 5 very easy)
Recommend to others (bespoke item) | 3 month follow-up
  The final item sought participants opinion on 'recommending the intervention to others. 'In your opinion, should we continue to offer this advice and information leaflets to other people attending our service? With three response options Yes/No/ Don't know

CONTACTS AND LOCATIONS:
Overall Officials: Corina Naughton, PhD, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Co Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual patient data (IPD) will be available on request from the authors Data will include participant demographics and outcome measures listed above
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From January 2024 for five years
Access Criteria: On request

REFERENCES:
- [Background] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Background] Ida S, Kaneko R, Murata K. SARC-F for Screening of Sarcopenia Among Older Adults: A Meta-analysis of Screening Test Accuracy. J Am Med Dir Assoc. 2018 Aug;19(8):685-689. doi: 10.1016/j.jamda.2018.04.001. Epub 2018 May 31. PMID 29778639
- [Background] Pearson E, Siskind D, Hubbard RE, Gordon EH, Coulson EJ, Warren N. Frailty and severe mental illness: A systematic review and narrative synthesis. J Psychiatr Res. 2022 Mar;147:166-175. doi: 10.1016/j.jpsychires.2022.01.014. Epub 2022 Jan 8. PMID 35051715
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Hays RD, Spritzer KL, Thompson WW, Cella D. U.S. General Population Estimate for "Excellent" to "Poor" Self-Rated Health Item. J Gen Intern Med. 2015 Oct;30(10):1511-6. doi: 10.1007/s11606-015-3290-x. Epub 2015 Apr 2. PMID 25832617
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Travers J, Romero-Ortuno R, Cooney MT. Testing the feasibility of a primary-care exercise intervention to prevent and reverse early frailty and build resilience in community-dwelling older adults. EClinicalMedicine. 2022 Mar 22;46:101355. doi: 10.1016/j.eclinm.2022.101355. eCollection 2022 Apr. PMID 35340628
- [Background] PROMIS (2021) GLOBAL HEALTH SCORING. MANUALhttps://www.healthmeasures.net/images/PROMIS/manuals/Scoring_Manual_Only/PROMIS_Global_Health_Scoring_Manual.pdf
- [Background] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT06127680/Prot_SAP_ICF_000.pdf